CLINICAL TRIAL: NCT03378492
Title: Utilizing Ultrasound for Residents as an Aid in Epidural Placement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not enroll, was closed
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2000021722
Record Dates: First submitted 2017-12-12; First posted 2017-12-19 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Epidural Placement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Epidural (Active Comparator): Participants in this group will have epidurals placed using standard practice.
  Interventions: Procedure: Standard Epidural
- Ultrasound Guided Epidural (Experimental): Participants in this group will have epidurals placed using standard practice with the assistance of ultrasound.
  Interventions: Device: Ultrasound Guided Epidural

INTERVENTIONS:
Device: Ultrasound Guided Epidural — Sterile ultrasound gel will be applied to the patient's back and the sterile device will be used to image the lumbar vertebrae in the area of the palpation-derived location. When the device is placed above the vertebral interspace, the 3D image mode will identify the spine midline and the depth from the skin to the epidural space. A single 3D ultrasound video loop of the vertebral interspace will be saved to confirm correct landmark identification. After identification of the vertebral interspace, the skin will be marked with a marking utensil or physical indentation at the point of needle entry indicated by the device. The epidural needle will then be placed in the same fashion as in the standard procedure group. The depth of the epidural needle placement will be measured and recorded following observation of loss of resistance.
  Arms: Ultrasound Guided Epidural
Procedure: Standard Epidural — The point of needle entry will be located using the landmarks technique. The specific level of epidural placement will be determined on a per-patient basis at the anesthesiologist's discretion. The spine midline will also be palpated to determine the approximate location of an interlaminar space. The needle will then be inserted at the appropriate location determined by the landmarks technique, and successful epidural placement will be confirmed by observation of loss of resistance and follow-up confirmation of analgesia. The depth of the epidural needle placement will be measured and recorded following observation of loss of resistance. The epidural catheter will be inserted and the procedure will continue according to the standard of care.
  Arms: Standard Epidural

SUMMARY:
This randomized controlled trial will evaluate the use of ultrasound as an aid for epidural placement in residents performing all epidural techniques under direct staff anesthesiologist supervision.

DETAILED DESCRIPTION:
The purpose of this study is to assess the abilities of the "Accuro" to assist in lumbar epidural placement in patients. It is hypothesized that the use of the Accuro will result in an increase of first-attempt success rates, defined as successful epidural needle placement on the first needle insertion attempt.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for vaginal delivery
* ASA-1, ASA-2, and ASA-3
* Patients with no known back deformities
* Ability to sit upright for epidural placement
* No prior lumbar surgery
* No allergies to ultrasound gel
* Pre-pregnancy BMI >= 30

Exclusion Criteria:

* Patients < 18 years of age

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Success Rate | Baseline (at time of procedure)
  Success rates are defined as successful epidural administration on the first needle insertion attempt. This outcome will be a dichotomous (yes/no) outcome.

SECONDARY OUTCOMES:
Needle passes | Baseline (at time of procedure)
  A needle pass is defined as any forward advancement or withdraw and forward redirection of the needle without withdraw from the skin. This outcome will capture the number of passes.
Needle insertion attempts | Baseline (at time of procedure)
  The number of needle insertion attempts is defined as advancement of the needle through the skin in an effort to enter the epidural space; a needle requiring withdrawal from the skin for reinsertion is to be counted as an additional insertion attempt.
Accuracy of needle insertion | Baseline (at time of procedure)
  The accuracy of needle insertion location is determined by the need to redirect (different angle) or reinsert the needle (different skin puncture site). This outcome will describe qualitatively the accuracy of the needle placement.
Vertebral level of epidural placement | Baseline (at time of procedure)
  Vertebral level of epidural placement is a record of the vertebral level where the epidural is administered. This will be confirmed via ultrasound imaging in both standard group and ultrasound group following epidural administration.
Time to landmark identification | Baseline (at time of procedure)
  Time to landmark identification is defined as the time interval between the start of needle puncture site identification and the time to first needle puncture attempt. The start time of needle puncture site identification in both the standard group and ultrasound group corresponds to when the resident physician first places his/her hand on the patient to palpate the back.
Time to loss of resistance | Baseline (at time of procedure)
  Time to loss of resistance is defined as the time interval between the first needle puncture attempt and the observation of loss of resistance.
Time to complete epidural analgesia administration | Baseline (at time of procedure)
  Time to complete epidural analgesia administration is defined as the time interval between the observation of loss of resistance and administration of analgesics through the epidural catheter.
Total technical procedure time | Baseline (at time of procedure)
  Total technical procedure time is defined as the sum of (iv) Time to landmark identification, (v) Time to loss of resistance, and (vi) Time to complete epidural analgesia administration. This technical procedure time measure the time between first placing hands on the patient to the administration of analgesia.
Epidural space depth | Baseline (at time of procedure)
  Epidural space depth is the depth from the skin to the epidural space as measured in centimeters (accurate to 0.1 cm).
Pain | Baseline (at time of procedure)
  Pain during epidural administration: to be assessed after the completion of catheter insertion (verbal rating scale [VRS], 0-10, 0 = no pain, 10 = maximum pain).
Analgesia efficacy rate | Baseline (at time of procedure)
  Analgesia efficacy rate: defined as VRS <= 1 and absence of unilateral or failed block at 20 minutes after injection of the loading dose
Time to comfort | Baseline (at time of procedure)
  Time to comfort after administration of the loading dose will be recorded in minutes.
Patient satisfaction | Follow Up (Up to 1 day)
  Patient satisfaction with the epidural administration, assessed after the administration of the loading dose (scale 0-10, 0 = not satisfied, 10 = completely satisfied).

IPD SHARING:
Plan to Share IPD: Undecided